CLINICAL TRIAL: NCT01382186
Title: Veterans' Experiences Using Secure Messaging on MyHealtheVet
Brief Title: Veterans Experiences Using Secure Messaging
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: RRP 11-397
Record Dates: First submitted 2011-06-15; First posted 2011-06-27 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-10

CONDITIONS: Telemedicine
Keywords: Qualitative; User, Computer Interface; quantitative; survey; telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Purposive Sampling: Purposive sampling was used to identify a sample of 33 Veterans who have been Personally Authenticated for the SM feature on MHV. Participants were recruited from each site (Tampa, Boston). Women were purposively recruited to ensure females were represented in data findings.
- Random Sampling: Random sampling was used to conduct a quantitative survey with 819 veterans to explore their experiences using secure messaging.

SUMMARY:
Deployment of Secure Messaging (SM) in primary care and women's clinics throughout the Veteran Health System by 2011 was an implementation priority for the Secretary and Under Secretary for Health for FY11 under the VHA T21 initiative. Secure Messaging is in early phases of implementation, this eHealth tool requires thoughtful evaluation to promote the successful implementation and dissemination of this tool. The primary aim of this project is to describe Veterans' experiences when using the SM feature on MyHealtheVet (MHV). This project has local, VISN, and national impact on the implementation and sustainability of the SM feature on MHV through its qualitative and quantitative examination of users' experiences. Findings from this research explores why Veterans choose to, or not to, use the SM feature on MHV, identify facilitators and barriers, and examine if experiences differ by health literacy or computer literacy. In addition to the interview data, findings from the usability testing and the quantitative survey findings build knowledge about Veterans' experiences using the SM feature on MyHealtheVet. These data will inform systems improvements, educational approaches, and marketing strategies to increase adoption and long-term utilization among Veterans.

DETAILED DESCRIPTION:
Project Background:

Secure Messaging is a VHA implementation priority to improve Veteran access to care. Successful deployment of Secure Messaging will support improved access to care, and improved healthcare outcomes in the Veteran population. To support these initiatives, and the successful implementation of this health informatics tools in the VHA, this project is exploring Veterans' perspectives' about adopting Secure Messaging and their experiences using Secure Messaging to inform systems improvements, educational approaches, and marketing strategies.

Objectives:

The primary aim of this project is to describe Veterans' experiences when using the Secure Messaging feature on My HealtheVet (MHV). This research is designed to explore why Veterans choose to, or not to, use the Secure Messaging feature on MHV, identify facilitators and barriers, and examine if experiences differ by health literacy or computer literacy. In addition to the interview data, findings from the usability testing provide user data about Veterans' skills and patterns when using Secure Messaging. This study was extended to conduct a mail-in quantitative survey evaluation of Veterans experiences, preferences, purposes and perceived facilitators and barriers for using, or not using Secure Messaging.

Methods:

This is a prospective mixed-methods descriptive study.

In Phase One: A purposive sampling was used to identify the sample of Veterans who have been Personally Authenticated for the Secure Messaging feature on My HealtheVet. Participants were recruited from two sites (Tampa n=18, Boston n=15). Phase 1 data collection procedures included: (1) surveys; (2) In-person interviews; (3) usability testing; (4) Secure Messaging secondary data collection; and (5) telephone interviews to complete study objectives.

In Phase Two: Random sampling was used to collect mail-in survey data from up to 1,000 Veteran participants who have been personally authenticated to use secure messaging. Quantitative data will be summarized using descriptive statistics to describe sample characteristics, frequency counts and proportions.

Study Status: The project team has completed data collection and analysis for Phase 1 and 2. Team is currently working on publications for dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been Personally Authenticated for the SM feature on MHV and
* who use SM independent of other caregivers, and
* cognitive impairment that prevents use of a personal computer.

Exclusion Criteria:

* Unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans in Tampa and Boston who have been Personally Authenticated for the SM feature on MHV.
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jolie N. Haun, PhD MS BS, Principal Investigator — James A. Haley Veterans' Hospital, Tampa, FL
Locations (2):
- United States (2):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

REFERENCES:
- [Result] Haun JN, Lind JD, Shimada SL, Martin TL, Gosline RM, Antinori N, Stewart M, Simon SR. Evaluating user experiences of the secure messaging tool on the Veterans Affairs' patient portal system. J Med Internet Res. 2014 Mar 6;16(3):e75. doi: 10.2196/jmir.2976. PMID 24610454
- [Result] Haun J, Lind JD, Shimada SL, Simon SR. Secure Messaging as a tool to facilitate Veteran-provider communication. Annals of anthropological practice. 2013 Jan 1; 37(2):57-74.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Purposive Sampling | Random Sampling
Started | 33 | 819
Completed | 32 | 819
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants were Veterans registered for My HealtheVet and opted-in to use Secure Messaging in the Tampa FL and Boston MA areas.
Groups:
- Purposive Sampling; Random Sampling: Veterans registered for My HealtheVet and opted-in to use Secure Messaging from the Tampa, FL and Boston, MA areas.
- Total: Total of all reporting groups
Arm/Group | Purposive Sampling | Random Sampling | Total
Number analyzed (Participants) | 33 | 819 | 852
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12) | 62 (13) | 60.75 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 107 | 114
  Male | 26 | 712 | 738
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 45 | 47
  Not Hispanic or Latino | 28 | 706 | 734
  Unknown or Not Reported | 3 | 68 | 71
Region of Enrollment [Number; unit: participants]
  United States | 33 | 819 | 852
Number of particpants with greater than or equal to high school education [Number; unit: participants] | 33 | 817 | 850
Number of participants with annual income of $35,001 or more [Number; unit: participants] | 21 | 434 | 455

OUTCOME MEASURES:

1. Primary Outcome: Usability of Secure Messaging
Description: To determine ease of use and usefulness of secure messaging. Purposive sample of 33 participants were assessed for their ability to complete the following tasks: navigate to Secure Messaging, log-in to My HealtheVet and Secure Messaging, Set user preferences, check Secure Message inbox, open and send Secure Message, Open and read Secure Message attachment. Measured as: (1) able to complete task; (2) able to complete task with some difficulty; (3) not able to complete task.
Time Frame: baseline
Population: This user-testing method was conducted with the first purposive sample of 33 participants in phase 1 of the study. The random sample of 819 participants in phase 2 were not a part of the user-testing study method.
Measure: Number; unit: participants
Groups:
- Purposive Sampling: Able to Complete Task: Veterans in this arm were able to complete the task.
- Purposive Sampling: Able to Complete Task With Difficulty: Veterans in this arm were able to complete task with some difficulty.
- Purposive Sampling: Not Able to Complete Task: Veterans in this arm were not able to complete the task.
Arm/Group | Purposive Sampling: Able to Complete Task | Purposive Sampling: Able to Complete Task With Difficulty | Purposive Sampling: Not Able to Complete Task
Number analyzed (Participants) | 33 | 33 | 33
participants
  Navigate to My HealtheVet Site | 21 | 10 | 2
  Log in to site | 30 | 2 | 1
  Set "User Preferences" | 23 | 8 | 2
  Check inbox | 33 | 0 | 0
  Use links within Secure Messaging | 33 | 0 | 0
  Open Secure Message | 33 | 0 | 0
  Open attachment | 33 | 0 | 0
  Send secure message | 30 | 3 | 0
  Choose secure message recipients | 32 | 0 | 1
  Categorize message subject | 9 | 0 | 24
  Formulate subject header | 18 | 0 | 15
  Formulate a secure message | 33 | 0 | 0

2. Primary Outcome: Secure Messaging Use and Content Patterns
Description: Extraction of secure messages over a three-month time frame to examine message content type, including: general, tests, medication, and appointments.
Time Frame: 3 months
Population: This method of secondary data collection was conducted with the purposive sample of 33 Veterans in phase 1 of the study. The random sample of 819 Veteran survey respondents in phase 2 were not included in this method of data collection.
Measure: Number; unit: secure messages
Units Other Than Participants: number messages
Arm/Group | Purposive Sampling
Number analyzed (Participants) | 33
Number analyzed (number messages) | 66
secure messages
  General | 36
  Test | 1
  Appointment | 15
  Medication | 10
  Other: System Related not Content Related | 4

3. Primary Outcome: Frequency of Electronic Resource Use
Description: Mail surveys examine Veterans frequency of electronic resource use.
Time Frame: baseline
Population: This is a primary outcome for phase 2 of the study which was measured in random sample of 819 Veterans. The purposive sample of 33 Veterans from phase 1 was not included in this method of the study.
Measure: Number; unit: participants
Arm/Group | Random Sampling
Number analyzed (Participants) | 819
participants
  Everyday use of computer | 662
  Everyday use of internet | 653
  Use My HealtheVet "a few times a month or less" | 629
  Using secure messaging 6 months or longer | 499
  Use secure messaging at least once a year | 486
  Use secure messaging at least once a month | 131

4. Primary Outcome: Reasons for Using Secure Messaging Tool on My HealtheVet
Description: Participants reported reasons for Using Secure Messaging tool on My HealtheVet
Time Frame: baseline
Population: This is a primary outcome for phase 2 of the study which was measured in random sample of 819 Veterans registered for My HealtheVet and opted in to use Secure Messaging. The sample of 33 Veterans from phase 1 was not included in this method of the study.
Measure: Number; unit: participant
Arm/Group | Random Sampling
Number analyzed (Participants) | 819
participant
  Completing medication refills | 546
  Medication questions | 313
  Managing appointments | 343
  Test results | 350
  Health related questions | 340
  Sensitive health topics | 67

5. Primary Outcome: Benefits of Using Secure Messaging
Description: Veterans report benefits of using Secure Messaging
Time Frame: baseline
Population: as for outcome 4
Measure: Number; unit: participant
Arm/Group | Random Sampling
Number analyzed (Participants) | 819
participant
  Good communication tool | 619
  Saves time | 590
  Easy to use | 544

6. Primary Outcome: Intention to Use Secure Messaging in the Future
Description: Veteran respondent intention to use Secure Messaging in the future
Time Frame: baseline
Population: as for outcome 4
Measure: Number; unit: participant
Arm/Group | Random Sampling
Number analyzed (Participants) | 819
participant | 689

7. Primary Outcome: Veterans That Believed Improvements to the Secure Messaging System Would Make the Tool More Useful in the Future Are Presented in the Table.
Description: Veterans were asked to report if improvements to the secure messaging system would make the tool more useful for use in the future.
Time Frame: baseline
Population: as for outcome 4
Measure: Number; unit: participant
Arm/Group | Random Sampling
Number analyzed (Participants) | 819
participant | 342

8. Primary Outcome: Veteran Need for Education Support for My HealtheVet and Secure Messaging Use.
Description: Veterans were asked to report if they would like to have education and support using My HealtheVet and the Secure Messaging tool.
Time Frame: baseline
Population: as for outcome 4
Measure: Number; unit: participant
Arm/Group | Random Sampling
Number analyzed (Participants) | 819
participant
  Reported need for education and support | 328
  Report Veterans would benefit from education | 652

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Purposive Sampling; Random Sampling: Serious and other [non-serious] adverse events were not collected/assessed.
Arm/Group | Purposive Sampling | Random Sampling
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes